CLINICAL TRIAL: NCT01708252
Title: Feasibility Study: Evaluation of the Ulthera® System for Obtaining Lift and Tightening of the Neck in Post-Surgery and Surgery Naive Patients Who Failed to Respond to a Previous Ultherapy™ Treatment
Brief Title: Feasibility Study: Treatment of Post-surgery and Surgery Naive Patients Who Failed to Respond to a Previous Ulthera Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ULT-127
Record Dates: First submitted 2011-11-07; First posted 2012-10-16 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2013-06

CONDITIONS: Skin Laxity
Keywords: Ulthera® System; Ultherapy™ Treatment; Ulthera, Inc.; Ultrasound treatment for skin tightening
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ulthera treatment group (Experimental): All subjects will receive an Ulthera System Treatment
  Interventions: Device: Ulthera System Treatment

INTERVENTIONS:
Device: Ulthera System Treatment — Focused ultrasound energy delivered below the surface of the skin
  Other Names: Ultherapy™

SUMMARY:
Up to 10 subjects will be enrolled. All subjects will receive an increased density UltherapyTM treatment at dual depth. Treatments will be provided to the lower 2/3 of the face and neck. Follow-up visits will occur at 90 and 180 days post-treatment. Study images will be obtained pre-treatment, 30-60 min post-treatment, and at each follow-up visit.

DETAILED DESCRIPTION:
This is a prospective, single-site, non-randomized clinical trial efficacy of an additional Ultherapy™ treatment for subjects who were minimal or non-responders at Day 90 in a previous Ulthera clinical trial. Global Aesthetic Improvement Scale scores and patient satisfaction questionnaires will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 30 to 65 years.
* Subject in good health.
* BMI < 30.
* Skin laxity in the submental area as demonstrated by a grade II or III on the Knize scale for classification of cosmetic deformity of the cervicomental angle
* Previous participation in ULT-107, and adequate compliance with all treatment and follow-up visits. Groups (surgery or surgery naïve) will be designated based on group assigned in ULT-107).
* Have not had any concomitant surgical or skin tightening procedures since their Ultherapy™ treatment with ULT-107.

Exclusion Criteria:

* Pregnant, lactating, or are planning to become pregnant, and/or not using a reliable form of birth control.
* Presence of an active systemic or local skin disease that may affect wound healing.
* Severe solar elastosis.
* Excessive subcutaneous fat on the cheeks.
* Excessive skin laxity on the lower face and neck
* Significant scarring in areas to be treated.
* Open wounds or lesions in the area to be treated.
* Severe or cystic acne on the area to be treated

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Improvement in lower face and neck skin laxity | 90 days post-treatment
  Efficacy will be assessed using the 90-day images compared to baseline
Cervicomental angle | 90 days post-treatment
  Efficacy will be assessed using the 90-day images compared to baseline.

SECONDARY OUTCOMES:
Overall aesthetic improvement | 90 days post-treatment
  Principal Investigator and subject will complete a Global Aesthetic Improvement Scale at 90 days post-treatment.
Patient satisfaction | 90 days post-treatment
  Subjects will complete a Patient Satisfaction Questionnaire at 90 days post-treatment.
Pain Assessment | Treatment visit
  Subject assessment of pain will be obtained using a 10-point validated Numeric Rating Scale following completion of each depth of treatment.
Patient Satisfaction | 180 days post-treatment
  Subjects will complete a Patient Satisfaction Questionnaire at 180 days post-treatment.
Overall aesthetic improvement | 180 days post-treatment
  Principal Investigator and subject will complete a Global Aesthetic Improvement Scale at 180 days post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Dayan, MD, FACS, Principal Investigator — DeNova Research
Locations (1):
- DeNova Research, Chicago, Illinois, United States